CLINICAL TRIAL: NCT02487550
Title: DC Vaccine Therapy Combined With Cytokine-Induced Killer Cell in Treating
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, xiaodong li, Principal Investigator, The First People's Hospital of Changzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIKRC001
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Renal Neoplasma
Keywords: Renal neoplasma; CIK cells

ARMS (2):
- DC-CIK (Experimental): Patients receive autologous dendritic cells (DC) loaded with autologous tumor lysate (DC vaccine) by endermic injection and infusion of CIK cells.
  Interventions: Biological: DC-CIK
- IL-2/IFN-α (Other): Patients receive treatment of IL-2 or IFN-α.
  Interventions: Biological: IL-2/IFN-α

INTERVENTIONS:
Biological: DC-CIK — Patients with renal cell carcinoma will receive autologous dendritic cells loaded with autologous tumor lysate (dendritic cell vaccine) by venous infusion of CIK cells.
  Arms: DC-CIK
Biological: IL-2/IFN-α — Patients with renal cell carcinoma will receive IL-2/IFN-α by venous infusion.
  Arms: IL-2/IFN-α

SUMMARY:
The purpose of this study is to show if vaccination with autologous dendritic cells pulsed with tumor lysate in combination with Cytokine-Induced Killer Cell (CIK) can induce a measurable immune response in patients with renal cell carcinoma, and to evaluate the clinical effect of the regimen.

DETAILED DESCRIPTION:
The purpose of this study is to show if vaccination with autologous dendritic cells pulsed with tumor lysate in combination with Cytokine-Induced Killer Cell (CIK) can induce a measurable immune response in patients with renal cell carcinoma, and to evaluate the clinical effect of the regime.

Primary

1. Determine the clinical responses(objective response, progression-free survival, and overall survival) in patients with renal cell carcinoma treated with autologous dendritic cells (DC) loaded with autologous tumor lysate (DC vaccine) in combination with Cytokine-Induced Killer Cell (CIK).

Secondary

1. Determine cellular immune response response in terms of immuknow assay, and correlate immune response with objective clinical response in patients treated with this regimen.
2. Determine safety of multiple administrations of this regimens in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma
* Age: > 18
* WHO- ECOG Performance Status 0-1
* At least one measurable tumor lesions according to the RECIST criteria.
* Life expectancy more than 3 months
* Written informed consent

Exclusion Criteria:

* Patients with a history of any other neoplastic disease less than 5 years ago (excepting treated carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin).
* Patients with metastatic disease in the central nervous system (CNS).
* Patients with other significant illness including severe allergy, asthma, angina pectoris or congestive heart failure.
* Patients with acute or chronic infection including HIV.
* Patients who are pregnant or nursing.
* Patients who have received antineoplastic therapy including chemotherapy or immunotherapy less than 4 weeks before beginning the trial.
* Patients who receive corticosteroids or other immunosuppressive agents.
* Patients with active autoimmune diseases such as lupus erythematosus, rheumatoid arthritis or thyroiditis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2015-08; Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free time | 3 months
Overall-survival time | 3 months

SECONDARY OUTCOMES:
Objective tumor response | 3 months